CLINICAL TRIAL: NCT04416542
Title: Inspire Home Study: Utilization of Home Monitoring During Therapy Optimization in Patients With an Inspire Upper Airway Stimulation System (Comparison of Home Sleep Testing vs. In-lab Polysomnography Testing)
Acronym: HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2020-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): Subjects in this group will be implanted with the Inspire UAS system and will undergo a standard in-lab PSG titration study at approximately 3 months post-activation and a 2-night HST at approximately 6 months post-activation
- Home Monitoring (Active Comparator): Subjects who have undergone implant of the Inspire UAS System and are randomized to this group will undergo a 2-night HST at 3 months post-activation. Depending on the results of the 2-night HST, the subject will either (a) undergo a PSG titration at 5 months post-activation and a 2-night HST at 6 months post-activation OR (b) undergo only a 2-night HST at approximately 6 months post-activation
  Interventions: Diagnostic Test: Home Sleep Testing

INTERVENTIONS:
Diagnostic Test: Home Sleep Testing — Two-night Home Sleep Tests (HSTs) will be conducted using commercially available Home Sleep Test equipment. The HST will be ordered by the clinical center through a HIPAA compliant HST service that has been selected by the study sponsor.
  The HSTs will be scored and interpreted according to AASM Guidelines by board certified sleep physicians affiliated with the HST service. The HST will be scored using the 4% oxygen desaturation rule.
  Arms: Home Monitoring

SUMMARY:
Inspire intends to conduct this study to compare Apnea-Hypopnea Index (AHI), between the two randomization arms, at 6 months post-activation

DETAILED DESCRIPTION:
This study is a prospective, randomized, non-blinded, multi-center study of therapy optimization related to the Inspire UAS System (implanted in a commercial setting under current labeling).

Comparison of outcomes between two (2) groups of patients (both implanted with the Inspire UAS system) who undergo different post-implant care algorithms throughout follow-up, in order to determine whether home sleep monitoring may be used as a surrogate for an in-lab PSG titration in a sub-set of patients.

Subjects who have been identified as candidates for Inspire therapy (implant of the Inspire UAS system), according to commercial labeling, will be recruited to participate in the study.

A maximum of 100 subjects will be enrolled at up to 5 clinical centers. A total of 60 subjects will be randomized (1:1) to one of two study arms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 22 years of age;
2. Patient has been diagnosed with moderate to severe OSA, with a baseline (pre-implant) AHI ≥ 15 based on a qualified sleep study;
3. Patient has been implanted with the Inspire UAS System but not yet activated, or has been scheduled for implant of the Inspire UAS System;
4. Patient currently owns a SmartPhone and is willing and able to install and use SmartPhone apps (at no cost to patient);
5. Patient is willing to utilize study equipment at home including Home Sleep Test (HST) equipment, pulse oximetry equipment, and sleep tracking equipment in accordance with the study protocol;
6. Patient is willing and able to return for all follow-up study visits;
7. Patient is willing to be randomized and adhere to randomization allocation;
8. Patient is willing to and capable of providing informed consent.

Exclusion Criteria:

1. Patient has central + mixed apneas more than > 25% of the total AHI;
2. Patient currently uses adjunctive sleep therapy (eg. CPAP, oral appliance, positional therapy) and will not discontinue use of adjunctive therapy upon implant of the Inspire UAS System;
3. Patient is pregnant or plans to become pregnant;
4. Patient has a terminal illness with life expectancy < 12 months;
5. Any other reason the investigator deems that the patient is unfit for participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Comparison of Apnea-Hypopnea Index (AHI), between the two randomization arms | 6 months post-activation
  The AHI endpoint will be determined by performing three equivalency tests for the following: Absolute AHI and, change in AHI. All comparisons will be done on the treatment AHI at 6 months between the control group and the home monitoring group. The objective is to demonstrate the equivalence in AHI, change in AHI, and response rate between the two groups.

SECONDARY OUTCOMES:
Comparison of Epworth Sleepiness Scale (ESS), between the two randomization arms | 6 months post-activation
  The Epworth Sleepiness Scale (ESS) endpoint will be determined by performing an equivalence test for the ESS score at 6 months between the control group and the home monitoring group. The objective is to demonstrate ESS score to be equivalent between the two groups.
  H0: |x ̃_diff |>2 Ha: |x ̃_diff |≤2
  where x ̃_diff is the median of differences (location shift) in the ESS score between the two groups.
  As the ESS score at 6 months has been shown to be non-normally distributed in previous studies, a non-parametric Hodges-Lehmann test at a significance level of 0.05 will be used to determine the location shift and its confidence interval between the two groups. An equivalence margin between -2 and 2 will be used as this is the defined meaningful clinical difference based on the AASM guidelines8.
Comparison of Oxygen Desaturation Index (ODI), between the two randomization arms | 6 months post-activation
  The Oxygen Desaturation Index (ODI) endpoint will be determined by performing an equivalence test for the ODI score at 6 months between the control group and the home monitoring group. The objective is to demonstrate ODI score to be equivalent between the two groups.
  H0: |x ̃_diff |>15 Ha: |x ̃_diff |≤15 where x ̃_diff is the median of differences (location shift) in the ODI score between the two groups.
  As the ODI score at 6 months has been shown to be non-normally distributed in previous studies, a non-parametric Hodges-Lehmann test at a significance level of 0.05 will be used to determine the location shift and its confidence interval between the two groups. ODI is closely related to AHI and therefore an equivalence margin of -15 and 15 will be used.
Comparison of Therapy Usage (hours per week), between the two randomization arms | 6 months post-activation
  The therapy usage endpoint will be determined by performing an equivalence test for the average therapy usage at 6 months between the control group and the home monitoring group. The objective is to demonstrate therapy usage to be equivalent between the two groups.
  H0: |x ̃_diff |>0.5 hrs Ha: |x ̃_diff |≤0.5 hrs where x ̃_diff is the median of differences (location shift) in therapy usage between the two groups.
  As the treatment therapy usage at 6 months has been shown to be non-normally distributed in previous studies, a non-parametric Hodges-Lehmann test at a significance level of 0.05 will be used to determine the location shift and its confidence interval between the two groups. An equivalence margin between -0.5 and 0.5 hrs will be used as this is the defined meaningful clinical difference based on the AASM guidelines8.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kent D, Huyett P, Yu P, Roy A, Mehra R, Rundo JV, Stahl S, Manchanda S. Comparison of clinical pathways for hypoglossal nerve stimulation management: in-laboratory titration polysomnography vs home-based efficacy sleep testing. J Clin Sleep Med. 2023 Nov 1;19(11):1905-1912. doi: 10.5664/jcsm.10712. PMID 37421320